CLINICAL TRIAL: NCT05513417
Title: Digital Care Programs for Female Pelvic Health: a Large-scale, Multi-disorder, Observational Study
Brief Title: Digital Care Programs for Female Pelvic Health
Status: Enrolling by invitation | Type: Observational
Sponsor: Sword Health, SA (Industry)
Responsible Party: Sponsor
Other Study IDs: BL-OBS-PH-US-01
Record Dates: First submitted 2022-08-19; First posted 2022-08-24 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Floor Disorders; Pelvic Pain; Pelvic Organ Prolapse; Pelvic Floor Muscle Weakness; Pelvic Pain Syndrome
MeSH Terms: conditions — Pelvic Floor Disorders; Pelvic Pain; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: These programs will cover participants with pelvic floor conditions which significantly impact their quality of life, to the extent they seek specialised care in direct relation to these conditions.
  Interventions: Device: Bloom Pod

INTERVENTIONS:
Device: Bloom Pod — Pelvic floor program consisting of exercise performed while using the device, education and behavioural change

SUMMARY:
The purpose of this study is to create a research repository, composed of data collected in the course of digital care programs for pelvic health conditions by SWORD Health/Bloom to individuals undergoing those programs.

This will allow the investigators to observe the acceptance, engagement and outcomes of programs using this approach in the treatment of multiple pelvic health disorders.

DETAILED DESCRIPTION:
This patient registry was designed as a research repository, composed of data collected in the course of digital care programs for pelvic health conditions by SWORD Health/Bloom to individuals undergoing those programs.

This data will allow the researchers to:

1. Assess the adoption, engagement and feasibility of digital care programs for pelvic musculoskeletal disorders and pelvic health;
2. Assess the results of digital care programs and compare the costs with the benefits obtained;
3. Correlate the results with patient's demographic and clinical profiles;
4. Examine the impact of mental health and the behavioral modification components of Bloom's interventions on disease markers, comorbidities, and productivity;
5. Increase the knowledge on several pelvic musculoskeletal disorders, namely how they progress and respond to digital care programs;
6. Develop new or improved tools to assist clinicians in the management of these disorders and in helping people achieve better pelvic health

The primary outcome will be the evolution of the participant's condition along the program. Depending on the condition, primary and secondary outcome measures vary, but the registry will include, in all cases, a complete characterisation of the participant's pelvic health status, as well as the periodic assessment of: a) performance indicators (through condition-specific tests); b) patient-reported outcomes (obtained using internationally validated pathology-specific questionnaires); c) pain levels; d) compliance; e) patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Signs/symptoms consistent with an acute (<12 weeks) or chronic (>12 weeks) abdominopelvic condition without signs/symptoms indicating underlying disease states that require immediate referral for medical management OR recovering from pelvic surgery with indication from their surgeon to engage in a pelvic physical therapy program
* Able to understand study procedures and willing to provide informed consent.

Exclusion Criteria:

* Health condition (cardiac, respiratory, neurological, immune) condition incompatible with at least 20 minutes of light to moderate exercise if not cleared by a physician to engage in an exercise program
* Bone fractures or other musculoskeletal conditions in which mobilization of the segment or joint is contra-indicated
* Rapidly progressive and new in onset neurological complaints if not cleared by a physician to engage in an exercise program; or signs of acute, serious neurologic compromise
* Active cancer diagnosis or receiving treatment for cancer if not cleared by a physician to engage in an exercise program
* Signs/symptoms consistent with inflammatory bowel diseases (Crohn's, ulcerative colitis, etc.)
* Signs/symptoms consistent with an active pelvic infection
* Aphasia, dementia or any other psychiatric comorbidity that interferes with the use of the medical device
* Complicated or high-risk pregnancy
* Hemodynamic instability
* Significant trauma to the area of pain within the last 12 weeks and functional incapacity and not cleared by a physician to engage in an exercise program
* Surgery within the last 12 weeks and not cleared by a physician to engage in an exercise program

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: These programs will cover patients suffering from pain and/or activity limitations in relation to the pelvic musculoskeletal systems, including but not limited to, pain/limitations affecting neuromusculoskeletal, genitourinary, gastrointestinal, and reproductive systems in this region. The programs will also cover patients submitted to surgery for a given pelvic condition involving any of the aforementioned systems.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2032-08 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported symptom level | Baseline, and then at regular intervals (after 9, 15 and 30 sessions) after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Pain Numerical Rating Scale referring to the previous 7 days. Higher scores mean more symptoms.
Pelvic Floor Impact Questionnaire - short form 7 (PFIQ-7) | Baseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  The PFIQ-7 consists of 7 questions that need to be answered 3 times each considering symptoms related to the bladder or urine, vagina or pelvis, and bowel or rectum and their effect on function, social health, and mental health in the past 3 months. The responses for each question range from "not at all" (0) to "quite a bit" (3). To get scale scores, the mean of each of the 3 scales is individually calculated, which ranges from 0-3, this number is then multiplied by 100 and then divided by 3. The scale scores are then added together to get the total PFIQ-7 score, which ranges from 0-300. A lower score means there is a lesser effect on quality of life.

SECONDARY OUTCOMES:
Anxiety | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time common to all conditions measured through General Anxiety Disorder-7 (GAD-7) is a 7-item scale (scores 0-21). Higher scores mean higher anxiety levels.
Depression | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time common to all conditions measured through Patient Health Questionnaire-9 (PHQ-9), a 9-item scale (0-27). Higher scores mean higher depression levels.
Work productivity and absenteeism | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time common to all conditions measured through Work Productivity and Activity Impairment Questionnaire (WPAI) assessed by the sub-scores: WPAI overall (combining presenteeism and absenteeism), WPAI work (presenteeism), WPAI time (absenteeism) and WPAI activities (activities of daily living impairment) (scores 0-100%). Higher scores mean greater impairment.
Self-reported consumption of painkillers | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time common to all conditions measured through Self-reported consumption of painkillers (yes/no); Prescription drugs (yes/no); Opioids (yes/no)
Self-reported intent to seek additional healthcare services | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time common to all conditions measured through a numerical rating scale (0-100). Higher scores mean higher intent.
Self-reported fatigue (VAS) | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time common to all conditions measured through a 0-10 Visual Analogue Scale. Higher scores mean higher fatigue.
Self-reported symptom level (VAS) | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  Change over time common to all conditions measured through a 0-10 Visual Analogue Scale. Higher scores mean more symptoms.

OTHER OUTCOMES:
Sessions performed | Measured at the end of the program, an average of 10 weeks
  Number of total exercise sessions performed
Self-reported satisfaction | aseline, then 3, 5 and 10 weeks after program initiation, and then at 6, 12 and 24 months after enrolment
  measured through the Net Promoter Score question collected at end of program: "On a scale from 0 to 10, how likely are you to recommend SWORD's programs to a friend or family member?")
Total treatment time | Measured at the end of the program, an average of 10 weeks
  Number of minutes spent on exercise sessions (aggregated)
Average treatment time per week | Measured at the end of the program, an average of 10 weeks
  Average number of minutes spent on exercise per week

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Correia, PhD, Principal Investigator — Sword Health, Inc
Locations (1):
- Sword Health Inc, Draper, Utah, United States

IPD SHARING:
Plan to Share IPD: No